CLINICAL TRIAL: NCT06144892
Title: Comparing the Comfort and Effectiveness of Proactive Airway Management Therapy for Sleep Apnea
Brief Title: The Comfort of Proactive Sleep Apnea Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovaResp Technologies Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: comfort study
Record Dates: First submitted 2023-11-17; First posted 2023-11-22 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Sleep Apnea; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention first (Experimental): Patients will undergo proactive therapy first, followed by the buffer period, and finally the conventional APAP therapy.
  Interventions: Device: Proactive Therapy
- Control first (Experimental): Patients will undergo the conventional APAP therapy first, followed by the buffer period, and finally the proactive therapy.
  Interventions: Device: Proactive Therapy

INTERVENTIONS:
Device: Proactive Therapy — Uses AI to make predictions and preventions of future apneic events.

SUMMARY:
The goal of this clinical trial is to compare in OSA patients who regularly adhere to CPAP therapy. The main question[s] it aims to answer are:

* To assess if proactive therapy can effectively treat OSA with lower mean therapy pressure compared to conventional APAP therapy
* To compare user comfort between proactive therapy and conventional APAP therapy

Participants will undergo the conventional APAP therapy and the new proactive therapy.

Researchers will compare nights in which conventional APAP was used and nights in which proactive therapy was used to see if patients were treated with lower pressures and effectively.

DETAILED DESCRIPTION:
This is a blinded, randomised, crossover, study on patients diagnosed with obstructive sleep apnea who regularly adhere to APAP therapy. Data collection will span 23 consecutive nights for each participant. Participants will use a modified APAP device for 2 periods of 9 nights each, separated by 5 nights in which participants will use their personal APAP device. The modified APAP device is switchable between two therapy modes: a) proactive therapy, and b) conventional APAP therapy. Treatment for the 2 periods will be randomly assigned, with one period as the test period where the proactive therapy is used every night for 9 consecutive nights, and the other as the control period where their conventional APAP therapy (i.e., the participant's regular therapy but on the modified device) is used every night for 9 consecutive nights. Participants will be blinded to the therapy they are receiving during the test and control period. Data will be collected by the modified PAP device and at-home sleep apnea test ring.

ELIGIBILITY:
Inclusion Criteria:

* Must be a current CPAP user
* Must have used a PAP device for more than 4 months.
* Before the first night of the study, participant must be willing to lend their personal PAP device for inspection in order for the study coordinator to transfer their PAP therapy settings to one of our modified PAP devices.
* Must be willing to wear the sleep diagnostic ring throughout each night of the study for the entire study duration (i.e., the full 23 days).
* Must be willing to have their CPAP SD memory card analyzed to determine their mean pressure and excess leak rate history
* Must be free of flu-like illness or any upper tract infection symptoms at the time of data collection.

Exclusion Criteria:

* Subjects actively using bi-level PAP or require oxygen therapy.
* Inspection of the participant's CPAP SD card data shows that history of highly frequent excess leak during therapy. Exclusion due to high leak will be determined on a case-by-case basis.
* History of severe cardiovascular disease, including NYHA Class III or IV heart failure, CAD with angina, or MI/stroke within past 6 months.
* Subjects who are medically complicated or who are medically unstable (i.e., cancer, dementia, unstable cardiac or respiratory disease, or unstable psychiatric illness)
* Potential sleep apnea complications that in the opinion of the clinician may affect the health and safety of the participant.
* Inability or unwillingness of individual to give written informed consent.
* Neuromuscular disease, hypoglossal-nerve palsy, severe restrictive or obstructive pulmonary disease, moderate-to-severe pulmonary arterial hypertension, severe valvular heart disease, New York Heart Association class III or IV heart failure, recent myocardial infarction or severe cardiac arrhythmias (within the past 6 months), persistent uncontrolled hypertension despite medication use, active psychiatric disease, and coexisting non-respiratory sleep disorders that would confound functional sleep assessment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-25 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Mask pressure | 18 nights
  Calculated as the mean pressure throughout the night.

SECONDARY OUTCOMES:
Apnea-Hypopnea Index | 18 nights
  Calculated as the mean number of apnea and hypopnea events throughout the night, in events/hr.
Comfort score | 18 nights
  Questionnaire that measures comfort of therapy.
Sleepiness self-assessment | 18 nights
  Patients will be requested to fill out a questionnaire to help evaluate their sleepiness after the treatment period and control period

IPD SHARING:
Plan to Share IPD: No